CLINICAL TRIAL: NCT02586766
Title: University of Michigan Youth Violence Prevention Emergency Department Brief Intervention
Brief Title: University of Michigan Youth Violence Prevention Emergency Department Brief Intervention (Project Sync)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Rebecca Cunningham, Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 5U01CE001957-05 (NIH)
Record Dates: First submitted 2015-10-09; First posted 2015-10-26 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Violence
Keywords: Youth Violence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral: Project Sync (Experimental): Brief 30 minute on-on-one private motivation interviewing intervention during emergency department care
  Interventions: Behavioral: Project Sync
- Comparison Group (No Intervention): This group did not receive an intervention, but did receive an informational pamphlet of resources in the area (enhanced usual care).

INTERVENTIONS:
Behavioral: Project Sync — A 30 minute private on-on-one brief motivational interviewing intervention given during emergency department care. The goal of the intervention was to reduce and prevention youth violence using techniques to change behavior in a respectful, non-confrontational, and non-judgmental manner. This one-on one counseling approach emphasizes individual choice and responsibility and differentiates between future goals/values and current behavior
  Arms: Behavioral: Project Sync

SUMMARY:
The purpose of this study is to determine whether a brief motivational interviewing intervention given during emergency department care to 14-20 year olds seeking treatment, could reduce youth violence.

DETAILED DESCRIPTION:
This Emergency Department (ED) based study will test the effectiveness of a tailored therapist delivered motivational interviewing intervention, and an informational pamphlet control condition (IC) on reducing violence in 14-20 year olds who present to the Hurley Medical Center (HMC). Eligible adolescents at the Hurley Medical Center (HMC) emergency department (ED) (based on eligibility criteria) will complete a computerized online survey. The goal of the intervention was to examine ways to reduce and prevention youth violence using techniques to change behavior in a respectful, non-confrontational, and non-judgmental manner. This one-on one counseling approach emphasizes individual choice and responsibility and differentiates between future goals/values and current behavior. At 2-months following their ED visit, eligible adolescents (both from the intervention group and control group) will meet with a research assistant and self-administer an online computerized follow-up survey. An online survey tool will be used for baseline, follow up and post-test surveys. Participants will self-administer the survey at the time of follow up, post-test and baseline.

ELIGIBILITY:
Inclusion Criteria:

1. adolescents (ages 14-20) presenting to the Hurley Medical Center for a medical injury or illness (except exclusions noted below);
2. adolescents will the ability to provide informed assent/consent depending on age;
3. access to a parent or guardian in person or by telephone for parental consent for adolescents ages 14-17 (over 90% of adolescents had a parent/guardian present based on our prior work);
4. currently residing in the intervention or control area;

Exclusion Criteria:

1. adolescents who do not understand English;
2. prisoners;
3. adolescents with abnormal vital signs;
4. adolescents deemed unable to provide informed consent by Emergency Department or research staff (e.g., intoxication, mental incompetence);
5. adolescents treated in the Emergency Department for suicide attempts or sexual assault (because they present in high psychological distress requiring intensive attention and intervention by Emergency Department staff).

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 409 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
violence behaviors as assessed with the combined modified Conflict Tactic Scale and the Conflict in Adolescent Dating Relationships Inventory to measure both peer and partner violence | past 2 months

REFERENCES:
- [Derived] Carter PM, Walton MA, Zimmerman MA, Chermack ST, Roche JS, Cunningham RM. Efficacy of a Universal Brief Intervention for Violence Among Urban Emergency Department Youth. Acad Emerg Med. 2016 Sep;23(9):1061-70. doi: 10.1111/acem.13021. Epub 2016 Sep 7. PMID 27265097